CLINICAL TRIAL: NCT02258191
Title: Pilot Study Evaluating Feasibility and Benefits of Telemonitored NIV Treatment on COPD Patients
Acronym: eCOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: eCOPD 001
Record Dates: First submitted 2014-09-24; First posted 2014-10-07 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: COPD
Keywords: NIV; COPD; telemonitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIV treatment with telemonitoring (Active Comparator): telemonitoring is used to manage NIV treatment
  Interventions: Device: telemonitoring
- NIV treatment with sham telemonitoring (Sham Comparator): sham telemonitoring (data not used for NIV management)
  Interventions: Device: sham telemonitoring

INTERVENTIONS:
Device: telemonitoring
  Other Names: Easy Care online
  Arms: NIV treatment with telemonitoring
Device: sham telemonitoring
  Other Names: Easy Care online
  Arms: NIV treatment with sham telemonitoring

SUMMARY:
Pilot study evaluating feasibility and benefits of telemonitored NIV (noninvasive ventilation) treatment on COPD (chronic obstructive pulmonary disease) patients.

Multicentric Randomized Controlled Trial

Primary Objective:

To evaluate benefits of telemonitoring system, Easy Care Online (ECO), on NIV long term treatment efficacy and patient compliance

Secondary Objectives:

To determine predictive factors of COPD exacerbation in patients treated by NIV with ECO To carry out a health economic evaluation on telemonitoring benefits in COPD pts treated with NIV

ELIGIBILITY:
Inclusion Criteria:

* COPD patient already treated by NIV requiring therapy assessment in their routine care Follow-Up or
* COPD patient requiring de Novo NIV therapy according to routine care rules (NIV<12h)
* Patient requiring NIV therapy by S9 VPAP ST +/- oxygen therapy
* Patient willing to participate to the study
* Patient or attendant able to complete patient passport and to come to Follow-Up visits.

Exclusion Criteria:

* NIV therapy Failure during screening phase (intolerance, patient refusal, significant leaks, significant AHI or Oxymetry events)
* Hospitalization conducting to NIV discontinuation for at least 1 week during the screening phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Blood Gaz and nocturnal transcutaneous carbon dioxyde partial pressure (PtCO2) evolution | 12 months
Compliance evolution: mean duration usage (hour per day) | 12 months

SECONDARY OUTCOMES:
Non-Intentional leaks | 12 months
Peripheral oxygen saturation (SP02) | 12 months
Apnea Hypopnea Index (AHI) | 12 months
Oxygen desaturation Index (ODI) | 12 months
Time with peripheral oxygen saturation (SP02) < 90% | 12 months
St Georges Quality of Life questionnaire | 12 months
6 Minutes Walking Test (6MWT) | 12 months
The Body-Mass Index, Airflow Obstruction, Dyspnea, and Exercise Capacity - (BODE) Index | 12 months
Epworth Sleepiness Scale (ESS) | 12 months
% of patients with Ventilatory asynchronisms | 12 months
Mean Noninvasive Ventilation (NIV) use duration (hour/day) | 12 months
% of days with noninvasive Ventilation (NIV) use ≥ 4h/day | 12 months
% of days with noninvasive Ventilation (NIV) use < 4h/day | 12 months
% of days with no Noninvasive Ventilation (NIV) use | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thibaut Gentina, MD, Principal Investigator — Hôpital Privé la Louvière - Lille
Locations (1):
- Hôpital privé la Louvière, Lille, France